CLINICAL TRIAL: NCT01202799
Title: A Phase 1, Randomized, Single Center, Open-Label, Multiple-Dose, Three-Way Crossover Study to Evaluate the Pharmacokinetics, Bioavailability and Safety of PENNSAID Gel in Comparison With Sandoz 75 mg Diclofenac Sodium Delayed Release Tablet and PENNSAID (Diclofenac Sodium Topical Solution) in Healthy Volunteers
Brief Title: Pharmacokinetics, Bioavailability and Safety of PENNSAID® Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: COV05100070
Record Dates: First submitted 2010-09-07; First posted 2010-09-16 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Pain
Keywords: Pharmacokinetics; Healthy volunteers; PENNSAID; Topical NSAID; Diclofenac
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 2% w/w diclofenac sodium topical gel
  Interventions: Drug: 2% w/w diclofenac sodium topical gel
- Treatment B (Active Comparator)
  Interventions: Drug: 1.5% w/w diclofenac sodium topical solution
- Treatment C (Active Comparator)
  Interventions: Drug: 75 mg diclofenac sodium delayed release tablet

INTERVENTIONS:
Drug: 2% w/w diclofenac sodium topical gel — 2% w/w diclofenac sodium topical gel
  Arms: Treatment A
Drug: 1.5% w/w diclofenac sodium topical solution — 1.5% w/w diclofenac sodium topical solution
  Arms: Treatment B
Drug: 75 mg diclofenac sodium delayed release tablet — 75 mg diclofenac sodium delayed release tablet
  Arms: Treatment C

SUMMARY:
It is anticipated that PENNSAID Gel will minimize systemic exposure versus oral diclofenac administered twice a day (BID). In addition, PENNSAID Gel should result in greater subject convenience and compliance with a comparable bioavailability, safety and tolerability profile to that of the approved PENNSAID solution administered four times a day (QID).

DETAILED DESCRIPTION:
PENNSAID Gel is a new topical gel formulation of diclofenac sodium that is similar in composition to PENNSAID solution.

No clinical studies have been conducted using PENNSAID Gel. The current study will compare the pharmacokinetics, bioavailability, safety and tolerability of diclofenac after the topical application of PENNSAID Gel with the approved formulations of topical PENNSAID Solution and oral Sandoz 75 mg diclofenac sodium delayed release tablets in healthy subjects.

The efficacy profile of PENNSAID Gel is based on the known efficacy profile of PENNSAID solution. Support for the BID dosing regimen includes the higher concentration of diclofenac sodium in PENNSAID Gel (2.0%) compared to PENNSAID solution (1.5%). In addition, compared to PENNSAID solution, PENNSAID Gel is designed to have better penetration of diclofenac to allow for a reduction in the number of applications per day from four to two while maintaining effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* The eligibility of subjects to enter the study is based on meeting the inclusion criteria listed below:

  1. Signed and dated IRB approved consent before any protocol procedures are performed.
  2. Males or non-pregnant, non-lactating females, minimum 18 years of age and maximum of 55 years of age.
  3. Female subjects must be negative on a serum pregnancy test, be postmenopausal for at least 1 year, surgically sterile, or using an acceptable form of contraception for 30 days prior to dosing and for the duration of study participation.
  4. Subjects with a body mass index (BMI) ≥19 and ≤29 kg/m².
  5. The findings from the ECG interpretation must be within the normal range.
  6. Subjects whose health status is assessed by the investigator as "normal healthy" by required screening and check-in assessments.
  7. Subjects must be able to provide written consent and agree to comply with study requirements.

Exclusion Criteria:

* Subjects will be ineligible for the study if they meet any of the following criteria:

  1. Known hypersensitivity to diclofenac, aspirin [acetylsalicylic acid (ASA)] or any other NSAID, dimethyl sulfoxide (DMSO) or ethanol. This includes subjects exhibiting aspirin or other NSAID-induced symptoms, including bronchospasm, rhinitis, and urticaria or other NSAID-induced allergic symptoms.
  2. Pregnant or lactating women. Women of reproductive potential (and women <12 months after menopause) may not participate unless they have agreed to use an effective contraceptive method while on study.
  3. Evidence of any serious active infections, severe uncontrolled cardiac, renal, hepatic, pulmonary or other systemic disease, significant medical or psychiatric illness, known seropositivity to HIV, known unexplained vision changes, history of unexplained syncope, lightheadedness, high blood pressure, chronic hepatic conditions like hepatic porphyria or clinically significant laboratory findings that would, in the investigators judgment, make the subject inappropriate for the study.
  4. Documented (upper GI series or endoscopy) gastroduodenal ulcer or any GI bleeding (except hemorrhoidal) within the last 6 months prior to screening.
  5. Abnormal hepatic and renal functions; hematologic changes:

     * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)≥2.5 X ULN
     * Gamma-glutamyl transpeptidase (GGT) ≥3X ULN
     * Total bilirubin ≥1.5X ULN
     * Serum creatinine ≥1.5X ULN
     * Hemoglobin ≤LLN.
  6. Major surgery or previous damage to the study knee(s) at any time (eg. total knee replacement, damage/reconstruction of the anterior or posterior cruciate ligaments), or minor knee surgery (eg, cartilage repair, collateral ligament repair, arthroscopic debridement) to the study knee(s) within 1 year prior to screening.
  7. Administration of a sedative hypnotic medication for insomnia within 14 days prior to screening.
  8. Administration of anti-depressants, within 60 days prior to screening.
  9. Administration of another investigational drug within the previous 30 days prior to screening.
  10. Skin disorder that affects palms of the hands or the application site of the knee(s).
  11. History of chronic headaches.
  12. Documented history of alcohol or drug abuse within 1 year prior to the screening visit
  13. Subjects who have smoked or used nicotine-containing products within 6 months prior to Period 1 dosing.
  14. Subjects treated with systemic or local diclofenac within one month of study Day 1.
  15. Using artificial exposure, tanning beds, or self-tanning cream on knee area within 90 days of study start.
  16. Donation or significant loss of blood (480 mL or more) within 30 days of dosing.
  17. Previous participation in this study or participation in another clinical trial within 30 days prior screening.
  18. Noncompliance with the study protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The rate and extent of exposure of diclofenac will be assessed. | During each of the 3 periods, blood samples will be obtained on Day 1 and Day 8 at pre-dose and 1, 2, 3, 4, 6, 8 and 12 hours post-dose; on Days 2-7 at pre-dose; and on Days 9, 13 and 15 at approximately 8 AM.
  Summary statistics including the mean, standard deviation, coefficient of variation, geometric mean and geometric %CV will be calculated for all PK parameters by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Gutierrez, MD, Principal Investigator — Comprehensive Phase One ®
Locations (1):
- Comprehensive Phase One, Miramar, Florida, United States

REFERENCES:
- [Derived] Holt RJ, Taiwo T, Kent JD. Bioequivalence of diclofenac sodium 2% and 1.5% topical solutions relative to oral diclofenac sodium in healthy volunteers. Postgrad Med. 2015 Aug;127(6):581-90. doi: 10.1080/00325481.2015.1058689. Epub 2015 Jun 16. PMID 26077436